CLINICAL TRIAL: NCT05753358
Title: Total Worker Health for Wildland Firefighters
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Collaborators: Federal Emergency Management Agency (U.S. Federal Agency); National Fallen Firefighters Foundation (Unknown)
Responsible Party: Principal Investigator, Kerry Kuehl, Professor of Medicine, Section Chief, and Director of Human Performance Laboratory, Oregon Health and Science University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: EMW-2018-FP-00284
Record Dates: First submitted 2023-02-10; First posted 2023-03-03 (Actual); Last update posted 2023-03-03 (Actual); Status verified 2023-02

CONDITIONS: Health Behavior; Total Worker Health; Occupational Health
Keywords: Sleep Hygiene; Cardiovascular Disease; Firefighter; Wildland; Occupational Hazards; Occupational Safety; health promotion
MeSH Terms: conditions — Health Behavior; Sleep Hygiene; Cardiovascular Diseases

STUDY DESIGN:
Intervention Model Description: This mixed-methods project had three phases. The initial qualitative phase was assessing the needs of wildland firefighters across segments and geographic locations to identify and prioritize program components. During the first phase, we recruited firefighters and collected baseline data in order to assess their needs. The second phase was to build a comprehensive, engaging TWH program for those fighting wildfires. It needed to be accessible on smartphone, tablet or computer, and suitable for individual, group and classroom settings. The final, third phase was to evaluate the program with a prospective proof-of-concept, usability and effectiveness trial among all types of wildland firefighters in different geographic locations.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Needs Assessment and Total Worker Health Program (Experimental): The initial phase was a needs assessment for wildland firefighters across segments and geographic locations to identify and prioritize program components. During the first phase, we recruited firefighters and collected baseline data in order to assess their needs using surveys for quantitative data and interviews and focus groups for qualitative data. The total worker health program includes 14, 30-minute modules on health topics highlighted during the needs assessment phase. Participants completed the program either individually or as part of a group.
  Interventions: Other: Total Worker Health for Wildland Firefighters

INTERVENTIONS:
Other: Total Worker Health for Wildland Firefighters — The program is structured as 30-minute modules that can be done individually, with a partner, as a group or in a classroom setting. The six core modules are supplemented with eight elective modules. The program can be accessed on a smartphone, tablet or computer, and if needed can be downloaded as a pdf.

SUMMARY:
The overarching goal is to develop, refine and disseminate a comprehensive, easily accessible and effective Total Worker Health (TWH) program for wildland firefighters (WFF).

The term Total Worker Health® (TWH) (NIOSH) refers to the synergistic combination of 1) health promotion (e.g., healthy nutrition, exercise, restorative sleep), 2) worker safety issues, such as protective equipment and hazard control, merged with 3) work organization change to support and promote TWH.

ELIGIBILITY:
Inclusion Criteria:

* any firefighter attending an OHSU-led informational meeting

Exclusion Criteria:

* Firefighters planning to retire from fire fighting work within 12 months will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2020-02-24 (Actual); Primary Completion 2022-04-14 (Actual); Study Completion 2022-04-14 (Actual)

PRIMARY OUTCOMES:
Change in Cardiovascular Risk Knowledge | 0 weeks to 14 weeks
  Change in cardiovascular risk knowledge was assessed using this survey question: "I know my risk factors for cardiovascular disease.". This was measured using a seven-point Likert agreement scale (1 = strongly disagree to 7 = strongly agree).
Change in Physical Activity | 0 weeks to 14 weeks
  Change in physical activity was assessed using this survey question: "On average, I get 150 minutes of moderate physical activity per week (including your work).". This was measured using a seven-point Likert agreement scale (1 = strongly disagree to 7 = strongly agree).
Change in Supplement Knowledge | 0 weeks to 14 weeks
  Change in supplement knowledge was assessed using this survey question: "I need supplements to balance the additional nutritional needs of being a wildland firefighter.". This was measured using a seven-point Likert agreement scale (1 = strongly disagree to 7 = strongly agree).
Change in Hydration Knowledge | 0 weeks to 14 weeks
  Change in hydration knowledge was assessed using the survey questions: "Camelback systems are more effective for maintaining hydration than canteens." and "Dehydration begins to affect performance when fluid loss equals 2% of body weight.". Both were measured using a seven-point Likert agreement scale (1 = strongly disagree to 7 = strongly agree).
Change in Nutrition Knowledge | 0 weeks to 14 weeks
  Change in nutrition knowledge was assessed using the survey questions: "Carbohydrates are the primary fuel for moderate to intense physical activity." and "Protein is contained in many foods, including bread and rice.". This was measured using a seven-point Likert agreement scale (1 = strongly disagree to 7 = strongly agree).
Change in Alcohol Knowledge | 0 weeks to 14 weeks
  Change in alcohol knowledge was assessed using the survey questions: "I know the definition of binge drinking." and " Drinking alcohol increases my cancer risk.". This was measured using a seven-point Likert agreement scale (1 = strongly disagree to 7 = strongly agree).
Change in Sleep Knowledge | 0 weeks to 14 weeks
  Change in sleep knowledge was assessed using the survey questions: "Power naps (15 to 30 minutes) will restore alertness and reduce accidents." and "Staying awake for 24 hours is equivalent to having a blood alcohol level greater than 0.08, the legal limit." and "Getting less than 5 hours of sleep lowers testosterone levels equal to someone 10 years older.". Both were measured using a seven-point Likert agreement scale (1 = strongly disagree to 7 = strongly agree).
Change in Mental Health Behavior | 0 weeks to 14 weeks
  Change in mental health behavior was assessed using the survey questions: "I am able to bounce back from stressful events." and "In general, I manage stress in a healthy way.". This was measured using a seven-point Likert agreement scale (1 = strongly disagree to 7 = strongly agree).
Change in Blood Pressure Knowledge | 0 weeks to 14 weeks
  Change in blood pressure knowledge was assessed using this survey question: "I know my blood pressure.". This was measured using a seven-point Likert agreement scale (1 = strongly disagree to 7 = strongly agree).
Change In Nutrition Behavior | 0 weeks to 14 weeks
  Change in nutrition behavior was assessed using this survey question: "I intend to eat every 2 hours while doing arduous wildland firefighting.". This was measured using a seven-point Likert agreement scale (1 = strongly disagree to 7 = strongly agree).
Change in Cancer Risk Knowledge | 0 weeks to 14 weeks
  Change in cancer risk knowledge was assessed using this survey question: "I know my risk factors for cancer.". This was measured using a seven-point Likert agreement scale (1 = strongly disagree to 7 = strongly agree).
Change in Alcohol Behavior with Sleep | 0 weeks to 14 weeks
  Change in alcohol behavior was assessed using this survey question: "I use alcohol to get to sleep.". This was measured using a seven-point Likert agreement scale (1 = strongly disagree to 7 = strongly agree).
Change in Primary Care Behavior | 0 weeks to 14 weeks
  Change in primary care behavior was assessed using this survey question: "It is important for me to have a primary care physician.". This was measured using a seven-point Likert agreement scale (1 = strongly disagree to 7 = strongly agree).
Change in Physical Activity Perception | 0 weeks to 14 weeks
  Change in physical activity perception was assessed using this survey question: "I can get in shape two weeks before a wildland fire season.". This was measured using a seven-point Likert agreement scale (1 = strongly disagree to 7 = strongly agree).
Change in Mental Health Self Perception | 0 weeks to 14 weeks
  Change in mental health self perception was assessed using the survey questions: "I feel overwhelmed with my work." and "During the last month, I felt significantly depressed.". This was measured using a seven-point Likert agreement scale (1 = strongly disagree to 7 = strongly agree).
Change in Alcohol Cancer Risk Knowledge | 0 weeks to 14 weeks
  Change in alcohol cancer risk knowledge was assessed using this survey question: "Drinking alcohol increases my cancer risk.". This was measured using a seven-point Likert agreement scale (1 = strongly disagree to 7 = strongly agree).
Change in Alcohol Behavior | 0 weeks to 14 weeks
  Change in alcohol behavior was assessed using this survey question: "I am currently trying to moderate my drinking.". This was measured using a seven-point Likert agreement scale (1 = strongly disagree to 7 = strongly agree).
Change in Support Perception | 0 weeks to 14 weeks
  Change in support perception was assessed using this survey question: "I can rely on people at work to support me.". This was measured using a seven-point Likert agreement scale (1 = strongly disagree to 7 = strongly agree).
Change in Sleep Hygiene Behavior | 0 weeks to 14 weeks
  Change in sleep hygiene behavior was assessed using this survey question: "Before going to sleep, I wipe soot and ash from my skin.". This was measured using a seven-point Likert agreement scale (1 = strongly disagree to 7 = strongly agree).
Change in Cardiovascular Risk Behavior | 0 weeks to 14 weeks
  Change in cardiovascular risk behavior was assessed using this survey question: "I intend to keep track of my risks for cardiovascular disease.". This was measured using a seven-point Likert agreement scale (1 = strongly disagree to 7 = strongly agree).
Change in Physical Exam Behavior | 0 weeks to 14 weeks
  Change in physical exam behavior was assessed using this survey question: "I intend to get a physical exam once a year.". This was measured using a seven-point Likert agreement scale (1 = strongly disagree to 7 = strongly agree).
Change in Heat Illness Knowledge | 0 weeks to 14 weeks
  Change in heat illness knowledge was assessed using this survey question: "When feeling over heated, the first thing to do is stop working.". This was measured using a seven-point Likert agreement scale (1 = strongly disagree to 7 = strongly agree).
Change in Injury Knowledge | 0 weeks to 14 weeks
  Change in injury knowledge was assessed using this survey question: "On steep and rocky terrain, it is best to move quickly to reduce risk of injury.". This was measured using a seven-point Likert agreement scale (1 = strongly disagree to 7 = strongly agree).
Program Usability and Effectiveness | 14 weeks
  Program usability and effectiveness was assessed using the survey question: "During the program, the educational modules were valuable for improving my health." and "This program was easy to use." and "This was an efficient way to learn the material." and "I learned ways to improve my health." and "These topics should be part of our training." and "I would recommend this program to my co-workers.". This was measured using a seven-point Likert agreement scale (1 = strongly disagree to 7 = strongly agree).
Technology Used for Program | 14 weeks
  Technology used for program was assessed using the survey question: "I primarily used this program on:" The options were 1) Phone, 2) Tablet, 3) Computer, 4) Other. For other, space was provided for participants to write in their answer.
How the Program was Completed | 14 weeks
  How the program was completed was assessed using the survey question: "I primarily used this program on:" The options were 1) By myself, 2) With other firefighters, 3) With my family, 4) Other. For other, space was provided for participants to write in their answer.

SECONDARY OUTCOMES:
Change in Body Mass Index | 0 weeks to 14 weeks
  Change in body mass index was measured in kg/m2.

CONTACTS AND LOCATIONS:
Locations (1):
- Oregon Health & Science University, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Brook RD, Rajagopalan S, Pope CA 3rd, Brook JR, Bhatnagar A, Diez-Roux AV, Holguin F, Hong Y, Luepker RV, Mittleman MA, Peters A, Siscovick D, Smith SC Jr, Whitsel L, Kaufman JD; American Heart Association Council on Epidemiology and Prevention, Council on the Kidney in Cardiovascular Disease, and Council on Nutrition, Physical Activity and Metabolism. Particulate matter air pollution and cardiovascular disease: An update to the scientific statement from the American Heart Association. Circulation. 2010 Jun 1;121(21):2331-78. doi: 10.1161/CIR.0b013e3181dbece1. Epub 2010 May 10. PMID 20458016
- [Background] Fritschi L, Glass DC. Firefighters and cancer: where are we and where to now? Occup Environ Med. 2014 Aug;71(8):525-6. doi: 10.1136/oemed-2014-102230. Epub 2014 Jul 4. No abstract available. PMID 24996680
- [Background] Kales SN, Soteriades ES, Christophi CA, Christiani DC. Emergency duties and deaths from heart disease among firefighters in the United States. N Engl J Med. 2007 Mar 22;356(12):1207-15. doi: 10.1056/NEJMoa060357. PMID 17377158
- [Background] Walton SM, Conrad KM, Furner SE, Samo DG. Cause, type, and workers' compensation costs of injury to fire fighters. Am J Ind Med. 2003 Apr;43(4):454-8. doi: 10.1002/ajim.10200. PMID 12645102
- [Background] Semmens EO, Domitrovich J, Conway K, Noonan CW. A cross-sectional survey of occupational history as a wildland firefighter and health. Am J Ind Med. 2016 Apr;59(4):330-5. doi: 10.1002/ajim.22566. Epub 2016 Jan 21. PMID 26792645
- [Background] Britton C, Lynch CF, Ramirez M, Torner J, Buresh C, Peek-Asa C. Epidemiology of injuries to wildland firefighters. Am J Emerg Med. 2013 Feb;31(2):339-45. doi: 10.1016/j.ajem.2012.08.032. Epub 2012 Nov 15. PMID 23158597
- [Background] Vincent GE, Aisbett B, Hall SJ, Ferguson SA. Fighting fire and fatigue: sleep quantity and quality during multi-day wildfire suppression. Ergonomics. 2016 Jul;59(7):932-40. doi: 10.1080/00140139.2015.1105389. Epub 2015 Dec 18. PMID 26452576
- [Background] Clement S, Schauman O, Graham T, Maggioni F, Evans-Lacko S, Bezborodovs N, Morgan C, Rusch N, Brown JS, Thornicroft G. What is the impact of mental health-related stigma on help-seeking? A systematic review of quantitative and qualitative studies. Psychol Med. 2015 Jan;45(1):11-27. doi: 10.1017/S0033291714000129. Epub 2014 Feb 26. PMID 24569086
- [Background] Kuehl KS, Elliot DL, Goldberg L, MacKinnon DP, Vila BJ, Smith J, Miocevic M, O'Rourke HP, Valente MJ, DeFrancesco C, Sleigh A, McGinnis W. The safety and health improvement: enhancing law enforcement departments study: feasibility and findings. Front Public Health. 2014 May 8;2:38. doi: 10.3389/fpubh.2014.00038. eCollection 2014. PMID 24847475
- [Background] Kuehl KS, Elliot DL, MacKinnon DP, O'Rourke HP, DeFrancesco C, Miocevic M, Valente M, Sleigh A, Garg B, McGinnis W, Kuehl H. The SHIELD (Safety & Health Improvement: Enhancing Law Enforcement Departments) Study: Mixed Methods Longitudinal Findings. J Occup Environ Med. 2016 May;58(5):492-8. doi: 10.1097/JOM.0000000000000716. PMID 27158956
- [Background] Elliot DL, Goldberg L, Duncan TE, Kuehl KS, Moe EL, Breger RK, DeFrancesco CL, Ernst DB, Stevens VJ. The PHLAME firefighters' study: feasibility and findings. Am J Health Behav. 2004 Jan-Feb;28(1):13-23. doi: 10.5993/ajhb.28.1.2. PMID 14977155
- [Background] Elliot DL, Goldberg L, Kuehl KS, Moe EL, Breger RK, Pickering MA. The PHLAME (Promoting Healthy Lifestyles: Alternative Models' Effects) firefighter study: outcomes of two models of behavior change. J Occup Environ Med. 2007 Feb;49(2):204-13. doi: 10.1097/JOM.0b013e3180329a8d. PMID 17293760
- [Background] Robertson M, Henning R, Warren N, Nobrega S, Dove-Steinkamp M, Tibirica L, Bizarro A; CPH-NEW Research Team. The Intervention Design and Analysis Scorecard: a planning tool for participatory design of integrated health and safety interventions in the workplace. J Occup Environ Med. 2013 Dec;55(12 Suppl):S86-8. doi: 10.1097/JOM.0000000000000036. PMID 24284761
- [Background] Andajani-Sutjahjo S, Liew TCH, Smith JF, Esekielu I, Mason G, Tariu I. Engaging community volunteers in participatory action research in Tamaki community of Auckland, New Zealand. Health Promot Int. 2018 Apr 1;33(2):219-228. doi: 10.1093/heapro/daw057. PMID 27543931
- [Background] Elliot DL, Goldberg L, MacKinnon DP, Ranby KW, Kuehl KS, Moe EL. Empiric validation of a process for behavior change. Transl Behav Med. 2016 Sep;6(3):449-56. doi: 10.1007/s13142-015-0343-y. PMID 27528533
- [Background] Mabry L, Elliot DL, Mackinnon DP, Thoemmes F, Kuehl KS. Understanding the durability of a fire department wellness program. Am J Health Behav. 2013 Sep;37(5):693-702. doi: 10.5993/AJHB.37.5.13. PMID 23985292
- [Background] MacKinnon DP, Elliot DL, Thoemmes F, Kuehl KS, Moe EL, Goldberg L, Burrell GL, Ranby KW. Long-term effects of a worksite health promotion program for firefighters. Am J Health Behav. 2010 Nov-Dec;34(6):695-706. doi: 10.5993/ajhb.34.6.6. PMID 20604695
- [Background] von Elm E, Altman DG, Egger M, Pocock SJ, Gotzsche PC, Vandenbroucke JP; STROBE Initiative. The Strengthening the Reporting of Observational Studies in Epidemiology (STROBE) statement: guidelines for reporting observational studies. PLoS Med. 2007 Oct 16;4(10):e296. doi: 10.1371/journal.pmed.0040296. PMID 17941714
- [Background] Chen SY, Feng Z, Yi X. A general introduction to adjustment for multiple comparisons. J Thorac Dis. 2017 Jun;9(6):1725-1729. doi: 10.21037/jtd.2017.05.34. PMID 28740688
- [Derived] Kuehl K, Elliot D, DeFrancesco C, McGinnis W, Ek S, Garg B. A Web-Based Total Worker Health Intervention for Those Fighting Wildland Fires: Mixed Methods Development and Effectiveness Trial. J Med Internet Res. 2023 Oct 25;25:e47050. doi: 10.2196/47050. PMID 37878362
- See also: an open source, cloud-based, software that allows researchers to sort "cards" into different categories. — https://kardsort.com/
- See also: an open source, cloud-based, qualitative software — https://www.taguette.org/
- See also: subscription platform for e-learning course development — https://articulate.com/360